CLINICAL TRIAL: NCT04472117
Title: PREPARE: Patient Centered Perioperative Experience
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-287
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Minimally Invasive Surgery (MIS) Hysterectomy
Keywords: Patient education; Perioperative setting; PREPARE; Patient centeREd PerioperAtive expeRiencE; 20-287

STUDY DESIGN:
Intervention Model Description: There will be three phases in this study. Phase I will comprise 25 evaluable women (15 pre-operatively and a separate 10 post-operatively). The results of the pre-operative interviews will be closely monitored for data saturation and we may stop accrual earlier than the planned 15. Phase II will comprise 100 evaluable women. Phase III will comprise 100 evaluable women. All patients will undergo standard-of-care MIS hysterectomy, with standard follow-up with the addition of the interventions and randomization takes place here. Phase III participants will be deemed evaluable if they complete required surveys and if their charts contain sufficient information to determine their day-surgery status.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual care and usual care plus video (Experimental): Phase I (completed 3/31/2021): A sample of patients in phase I will complete a qualitative interview prior to or after surgery. Twenty-five evaluable patients (15 pre-operatively and a separate 10 post-operatively) will be selected to participate in an in-person/phone interview. Phase II: A separate group of women will compose phase II. All patients (N = 100) in phase II will complete discrete-choice surveys. Patients in phase III of the study will be randomized evenly to usual care plus video or usual care only. Phase III: One hundred participants will be randomized via CRDB to receive standard pre-operative counseling or standard pre-operative counseling with the additional of an educational video. Those randomized to view the video will also complete the post-video survey. All patients will complete the post-op survey.
  Interventions: Other: usual care; Other: Educational video

INTERVENTIONS:
Other: usual care — Interviews will be conducted in person or by telephone by an MD on the research team who does not have an ongoing treatment relationship with the patient, and has been trained by the qualitative methods specialist. Interviews will take place over the phone or in person and are anticipated to last approximately 20-30 minutes.
  Other Names: Qualitative Interviews
Other: Educational video — Watch an educational video created by the research team and.will also complete the post-video survey. Those randomized to view the video must complete the post-video survey (Appendix 3), and all patients must complete the Post-Op Survey with the Patient Experience and Decision Regret Scale (Appendix 5) to be evaluable. If not completed, they will be replaced.

SUMMARY:
The purpose of this study is to determine whether an educational video about patients' perioperative experience (period that spans from the time of admission to the hospital to the time of recovery after surgery) will affect the timing of hospital discharge. The researchers will use information collected during this study to create a questionnaire and an educational video related to the patient perioperative experience. The educational video will address patient concerns about the perioperative period and recovery after surgery (post-operative recovery).

All participants in this study will be undergoing a MIS hysterectomy according to their routine care in the Gynecology

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥18 years of age.
* Scheduled to undergo MIS hysterectomy by a gynecologic oncologist at MSK at either Josie Robertston Surgery Center or the main hospital OR completed MIS hysterectomy by a gynecologic oncologist at MSK at either Josie Robertson Surgery Center or the main hospital within 1 month of consent (post-op patients eligible for Phase 1 only). Phase 1 was completed on 3/31/2021).
* Determined to be an appropriate candidate for the AXR program or expected to be discharged within 23 hours after surgery.

Exclusion Criteria:

* Not able to speak and read English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman undergoing MIS hysterectomy
Enrollment: 300 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Percentages of Ambulatory Extended Recovery (AXR) vs same day discharge | 2 years

SECONDARY OUTCOMES:
Patient satisfaction | 2 years
  Data from the discrete-choice experiment will be used to summarize patients' preferences and priorities. The discrete-choice experiment will entail a series of 28 side-by-side comparisons of hypothetical scenarios.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Jewell, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm